CLINICAL TRIAL: NCT00330018
Title: An Investigator Initiated Prospective Randomized, Controlled Pilot Study in Order to Evaluate the Place of Valganciclovir in Prevention of Cytomegalovirus Reactivation Following Allogeneic Stem Cell Transplantation
Brief Title: Valganciclovir in Prevention of Cytomegalovirus (CMV) Reactivation Following Allogeneic-Stem Cell Transplantation (SCT)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Hadassah Medical Organization (Other)
Responsible Party: Michael Shapira, MD, Hadassah University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: MYS-03-HMO-CTIL
Record Dates: First submitted 2006-05-24; First posted 2006-05-25 (Estimated); Last update posted 2015-04-21 (Estimated); Status verified 2009-08

CONDITIONS: Bone Marrow Transplantation; Cytomegalovirus
Keywords: BMT; CMV; GVHD
MeSH Terms: interventions — Valganciclovir; Acyclovir

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): PO Valganciclovir
  Interventions: Drug: Valganciclovir
- 2 (Active Comparator): PO Acyclovir
  Interventions: Drug: Acyclovir

INTERVENTIONS:
Drug: Valganciclovir — Valganciclovir
  Arms: 1
Drug: Acyclovir — Acyclovir
  Arms: 2

SUMMARY:
The rationale for this protocol is based on the need to assess if the current post stem cell transplantation CMV prophylaxis strategies (e.g. high-dose acyclovir plus pre-emptive treatment) can be improved by the use of valganciclovir. CMV is the most common viral infection following stem cell transplantation, causing significant morbidity and mortality. Furthermore, CMV has been shown to be associated with a number of indirect effects in SCT recipients including allograft dysfunction, acute and chronic graft versus host disease (GVHD). Valganciclovir is shown to be more active than oral ganciclovir, and as good as intravenous (i.v.) ganciclovir in treating newly diagnosed CMV retinitis. The use of valganciclovir for CMV prophylaxis post stem cell transplantation was never tested in controlled study. The investigators therefore suggest a prospective, randomized study to evaluate the efficacy and safety of valganciclovir compared with acyclovir for prevention of CMV disease in allogeneic stem cell transplantation recipients.

DETAILED DESCRIPTION:
Cytomegalovirus (CMV), the most common viral infection following stem cell transplantation (SCT), causes significant morbidity and mortality. It can result in CMV pneumonitis, hepatitis, encephalitis and gastrointestinal disease, as well as fever and neutropenia. Furthermore, CMV has been shown to be associated with a number of indirect effects in SCT recipients including reduced long-term patient survival, increased risks of opportunistic infections, allograft dysfunction, acute and chronic graft vs. host disease (GVHD). SCT patients at highest risk are seronegative donors, matched unrelated donors, SCT with T-cell depletion, patients after cord blood SCT, and patients with GVHD.

Valganciclovir, a valine ester pro-drug of ganciclovir, was developed to overcome the limitations of oral and i.v. ganciclovir, with a single once-daily 900 mg oral dose providing comparable plasma ganciclovir exposures to those achieved with 5 mg/kg i.v. ganciclovir. Its bioavailability is up to 10-fold higher than that of oral ganciclovir (same as above). There is already extensive clinical experience with valganciclovir in AIDS patients, where it has proved as effective as i.v. ganciclovir in treating newly diagnosed CMV retinitis, and in patients after solid organ transplant but no comparative data exists in patients after SCT.

We therefore planned a prospective, randomized study to evaluate the efficacy and safety of valganciclovir compared with acyclovir for prevention of CMV disease in SCT recipients.

ELIGIBILITY:
Inclusion Criteria:

1. Undergoing allogeneic SCT from a matched related or unrelated donor without T cell depletion.
2. Had an acceptable engraftment.
3. Can take oral medications within 10 days of engraftment.
4. Either the recipient or donor (or both) is CMV seropositive.

Exclusion Criteria:

1. Not fulfilling the inclusion criteria.
2. History of CMV infection or disease.
3. Anti-CMV therapy within the past 15 days.
4. Severe, uncontrolled diarrhea.
5. Both recipient and donor are CMV seronegative.
6. Evidence of malabsorption.
7. Inability to comply with study requirements.
8. Known hypersensitivity or other contraindication to ganciclovir or valganciclovir.
9. Pregnant or lactating patients.

Ages: 14 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2006-02; Primary Completion 2010-04 (Actual); Study Completion 2010-04 (Actual)

PRIMARY OUTCOMES:
Prevention of CMV reactivation | 100d

SECONDARY OUTCOMES:
Occurrence of CMV disease | 6m
Overall survival | 6m
Occurrence of GVHD | 6m
Occurrence of other infections | 6m

CONTACTS AND LOCATIONS:
Overall Officials: Michael Y Shapira, MD, Principal Investigator — Hadassah Medical Organization
Locations (1):
- Hadassah Medical Organization,, Jerusalem, Israel